CLINICAL TRIAL: NCT04865289
Title: A Phase 3 Randomized, Open-Label, Study of Pembrolizumab (MK-3475) Plus Lenvatinib (E7080/MK-7902) Versus Chemotherapy for First-line Treatment of Advanced or Recurrent Endometrial Carcinoma (LEAP-001)
Brief Title: Pembrolizumab (MK-3475) Plus Lenvatinib (E7080/MK-7902) Versus Chemotherapy for Endometrial Carcinoma (ENGOT-en9 / MK-7902-001) - China Extension Study
Acronym: LEAP-001
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7902-001 China Extension; MK-7902-001 (Other: MSD); ENGOT-en9 (Other: European Network for Gynaecological Oncological Trial groups); 194710 (Registry Identifier: JAPIC-CTI); 2023-505614-17 (Other: EU CT)
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Results first posted 2024-10-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Endometrial Neoplasms
MeSH Terms: conditions — Endometrial Neoplasms | interventions — lenvatinib; pembrolizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lenvatinib + Pembrolizumab (Experimental): Participants receive lenvatinib daily and pembrolizumab once at the start of each 3-week treatment cycle.
  Interventions: Drug: Lenvatinib; Biological: Pembrolizumab
- Paclitaxel + Carboplatin (Active Comparator): Participants receive paclitaxel and carboplatin once at the start of each 3-week treatment cycle.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib 4 mg or 10 mg capsules at a total daily dose of 20 mg taken by mouth once per day.
  Other Names: E7080, MK-7902, LENVIMA®
  Arms: Lenvatinib + Pembrolizumab
Biological: Pembrolizumab — Pembrolizumab 200 mg IV infusion given on Day 1 of each cycle.
  Other Names: MK-3475, KEYTRUDA®
  Arms: Lenvatinib + Pembrolizumab
Drug: Paclitaxel — Paclitaxel 175 mg/m^2 IV infusion given on Day 1 of each cycle.
  Other Names: TAXOL®, ONXAL®
  Arms: Paclitaxel + Carboplatin
Drug: Carboplatin — Carboplatin 10 mg/mL IV infusion at a total dose of are-under-the-curve (AUC) 6 (per Calvert's formula) given on Day 1 of each cycle.
  Other Names: PARAPLATIN®
  Arms: Paclitaxel + Carboplatin

SUMMARY:
The purpose of this study is to compare the efficacy of pembrolizumab + lenvatinib to chemotherapy in female participants with Stage III, IV, or recurrent endometrial carcinoma. It is hypothesized that the combination of pembrolizumab + lenvatinib will be superior to chemotherapy for progression-free survival (PFS) per Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) by blinded independent central review (BICR). It is also hypothesized that the combination of pembrolizumab + lenvatinib will be superior to chemotherapy for overall survival (OS).

As of Amendment 7 eligible participants on study completion will be able to transition to an extension study, if available, in which they can continue to receive pembrolizumab monotherapy, lenvatinib monotherapy, or a combination of both pembrolizumab and lenvatinib as received in the parent study.

DETAILED DESCRIPTION:
This China extension study will include participants previously enrolled in China in the global study for MK-7902-001 (NCT03884101) plus those enrolled during the China extension enrollment period.

ELIGIBILITY:
Inclusion Criteria:

* Has Stage III, Stage IV, or recurrent, histologically-confirmed endometrial carcinoma with disease that is either measurable or nonmeasurable but radiographically apparent, per RECIST 1.1 as assessed by BICR (note: may have received prior chemotherapy only if administered concurrently with radiation; may have received prior radiation without concurrent chemotherapy; may have received prior hormonal therapy for treatment of endometrial carcinoma, provided that it was discontinued ≥1 week prior to randomization; and may have received 1 prior line of systemic platinum-based adjuvant and/or neoadjuvant chemotherapy)
* Has provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion that was not previously irradiated, for determination of mismatch repair (MMR) status
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, as assessed within 7 days prior to the first dose of study intervention
* Is not pregnant or breastfeeding, and is either not a woman of childbearing potential (WOCBP) or is a WOCBP who agrees to use contraception during the study and for ≥120 days after pembrolizumab, ≥30 days after lenvatinib, or ≥180 days after (chemotherapy) [if a WOCBP, a pregnancy test will be required within 24 hours of first dose of study drug]
* Has adequately controlled blood pressure within 7 days prior to randomization
* Has adequate organ function based on assessment within 7 days prior to the first dose of study intervention

Exclusion Criteria:

* Has carcinosarcoma (malignant mixed Műllerian tumor), endometrial leiomyosarcoma or other high grade sarcomas, or endometrial stromal sarcomas
* Has a central nervous system (CNS) metastasis, unless local therapy (e.g., whole brain radiation therapy, surgery, or radiosurgery) has been completed and have discontinued use of corticosteroids for this indication for ≥4 weeks prior to starting study medication (major surgery within 3 weeks of the first dose of study drug will be exclusionary)
* Has a known additional malignancy (other than endometrial carcinoma) that is progressing or has required active treatment in the last 3 years
* Has gastrointestinal malabsorption or any other condition that might affect the absorption of lenvatinib
* Has a pre-existing Grade ≥3 gastrointestinal or nongastrointestinal fistula
* Has radiographic evidence of major blood vessel invasion/infiltration
* Has active hemoptysis (bright red blood of ≥0.5 teaspoon) within 3 weeks prior to the first dose of study intervention, or tumor bleeding within 2 weeks prior to randomization
* Has clinically significant cardiovascular disease within 12 months from first dose of study intervention including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability
* Has any infection requiring systemic treatment
* Has not recovered adequately from any toxicity and/or complications from major surgery prior to randomization
* Has a known history of human immunodeficiency virus (HIV) infection (HIV test is required at screening)
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (hepatitis B and C testing is required at screening)
* Has a history of (noninfectious) pneumonitis that required treatment with steroids, or has current pneumonitis
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to randomization
* Has an active autoimmune disease (with the exception of psoriasis) that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs)
* Has received prior systemic chemotherapy in any setting for the treatment of endometrial carcinoma (note: prior chemotherapy administered concurrently with radiation is permitted)
* Has received prior radiotherapy within 4 weeks prior to randomization (participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis - a 2-week washout is permitted for palliative radiation to non-CNS disease and vaginal brachytherapy)
* Has received prior hormonal therapy for the treatment of endometrial carcinoma within 1 week of randomization
* Has received prior therapy with any treatment targeting vascular endothelial growth factor (VEGF)-directed angiogenesis, an anti-programmed cell death (PD)-1, anti-PD ligand (L)1, or anti-PD L2 agent, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137)
* Has received a live or live attenuated vaccine within 30 days prior to the first dose of study intervention
* Has known intolerance to study intervention (or any of the excipients)
* Has had an allogenic tissue/solid organ transplant
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2025-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (22):
- China (22):
  - Anhui Cancer Hospital-Gynecological Oncology ( Site 2509), Hefei, Anhui
  - Beijing Obstetrics and Gynecology Hospital Capital Medical University ( Site 2505), Beijing, Beijing Municipality
  - Peking Union Medical College Hospital ( Site 2501), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 2504), Beijing, Beijing Municipality
  - Chongqing Cancer Hospital ( Site 2513), Chongqing, Chongqing Municipality
  - The First Affiliated hospital of Xiamen University-Obstetrics and gynecology department ( Site 2522), Xiamen, Fujian
  - The First Affiliated Hospital.Sun Yat-sen University ( Site 2507), Guangzhou, Guangdong
  - Guang Xi Tumour Hospital, Department of Chemotherapy ( Site 2517), Nanning, Guangxi
  - Harbin Medical University Cancer Hospital ( Site 2520), Harbin, Heilongjiang
  - Hubei Cancer Hospital ( Site 2510), Wuhan, Hubei
  - Xiangya Hospital Central-South University ( Site 2512), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 2523), Changsha, Hunan
  - Nanjing Maternity and Child Health Care Hospital ( Site 2508), Nanjing, Jiangsu
  - Jiangxi Maternal and Child Health Hospital ( Site 2519), Nanchang, Jiangxi
  - The First Hospital Of Jilin University ( Site 2518), Changchun, Jilin
  - The first affiliated Hospital of Xi an Jiaotong University ( Site 2502), Xi'an, Shaanxi
  - Fudan University Shanghai Cancer Center ( Site 2500), Shanghai, Shanghai Municipality
  - Obstetrics and Gynecology Hosp. Fudan University ( Site 2503), Shanghai, Shanghai Municipality
  - Shanghai First Maternity and Infant Hospital ( Site 2524), Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xinjiang Medical University ( Site 2515), Ürümqi, Xinjiang
  - Women s Hospital School of Medicine Zhejiang University ( Site 2511), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 2506), Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 130 participants were enrolled in China. 66 participants were randomized in the global portion for MK-7902-001 (NCT03884101) and 64 in the China extension portion.
Groups:
- Lenvatinib + Pembrolizumab: Participants received lenvatinib daily and pembrolizumab once at the start of each 3-week treatment cycle.
- Paclitaxel + Carboplatin: Participants received paclitaxel and carboplatin once at the start of each 3-week treatment cycle.
Period: Overall Study
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Started | 74 | 56
Treated | 73 | 56
Completed | 0 | 0
Not Completed | 74 | 56
Not completed — Death | 34 | 25
Not completed — Physician Decision | 27 | 27
Not completed — Sponsor Decision | 11 | 1
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Population: All Chinese participants who were randomized to the global study (NCT03884101) and to the extension portion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin | Total
Number analyzed (Participants) | 74 | 56 | 130
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (8.1) | 58.3 (7.3) | 60.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 56 | 130
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 74 | 55 | 129
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 74 | 56 | 130
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Participants were stratified by an ECOG Performance Status of 0 (Fully active, able to carry on all pre-disease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature).
  Participants
    ECOG = 0 | 35 | 29 | 64
    ECOG = 1 | 39 | 27 | 66
Prior Chemotherapy and/or Chemoradiation [Count of Participants; unit: Participants] — Participants were stratified by whether or not they had received prior chemotherapy and/or chemoradiation treatment; yes or no.
  Participants
    Yes | 21 | 18 | 39
    No | 53 | 38 | 91
Mismatch Repair (MMR) Status [Count of Participants; unit: Participants] — Participants were stratified by their MMR status; Mismatch Repair Proficient (pMMR) or Mismatch Repair Deficient (dMMR).
  Participants
    dMMR | 17 | 12 | 29
    pMMR | 57 | 44 | 101

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in Mismatch Repair Proficient (pMMR) Participants
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The PFS of pMMR participants was presented.
Time Frame: Up to approximately 45 months
Population: All pMMR Chinese participants who were randomized to the global study (NCT03884101) and to the extension portion were analyzed according to the treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 57 | 44
Months | 10.3 [6.4 to 12.7] | 10.2 [8.3 to 10.6]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Other — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.51 to 1.41]

2. Primary Outcome: PFS Based on RECIST 1.1 as Assessed by BICR in All Randomized Participants
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The PFS of all randomized participants was presented.
Time Frame: Up to approximately 45 months
Population: All Chinese participants who were randomized to the global study (NCT03884101) and to the extension portion were analyzed according to the treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 74 | 56
Months | 11.7 [8.3 to 19.4] | 10.3 [8.3 to 12.5]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Other — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.48 to 1.21]

3. Primary Outcome: Overall Survival (OS) in pMMR Participants
Description: OS was measured from the time of randomization up to death due to any cause. Participants without documented death at the time of the final analysis were to be censored at the date of the last follow-up. The OS for pMMR participants is presented.
Time Frame: Up to approximately 45 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 57 | 44
Months | 37.1 [19.5 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [21.7 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Non-Inferiority — The null hypothesis for the non-inferiority test was that the hazard ratio was equal to 1.1; p = 0.5831415, Log Rank; One-sided p-value based on log-rank test; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.64 to 2.15] — Based on Cox regression model with Efron's method for tie handling with treatment as a covariate
Statistical Analysis 2: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Superiority; p = 0.6980186, Log Rank; One-sided p-value based on log-rank test; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.64 to 2.15] — Based on Cox regression model with Efron's method for tie handling with treatment as a covariate

4. Primary Outcome: OS in All Randomized Participants
Description: OS was measured from the time of randomization up to death due to any cause. Participants without documented death at the time of the final analysis were to be censored at the date of the last follow-up. The OS for all randomized participants is presented.
Time Frame: Up to approximately 45 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 74 | 56
Months | NA [29.8 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [25.1 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Superiority; p = 0.52046, Log Rank; One-sided p-value based on log-rank test; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.57 to 1.80] — Based on Cox regression model with Efron's method for tie handling with treatment as a covariate

5. Secondary Outcome: Objective Response Rate (ORR) Based on RECIST 1.1 as Assessed by BICR in pMMR Participants
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1. The percentage of pMMR participants who experienced a CR or PR is presented.
Time Frame: Up to approximately 45 months
Population: Per the statistical analysis plan, all pMMR Chinese participants who were randomized to the global study (NCT03884101) and to the extension portion with measurable disease at the baseline scan were analyzed according to the treatment arm to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 55 | 44
Percentage of Participants | 50.9 [37.1 to 64.6] | 61.4 [45.5 to 75.6]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Other; p = 0.8497, Miettinen & Nurminen; One sided p value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentage = -10.5, 95% CI 2-sided [-29.2 to 9.3]

6. Secondary Outcome: ORR Based on RECIST 1.1 as Assessed by BICR in All Randomized Participants
Description: ORR was defined as the percentage of participants who had a CR: Disappearance of all target lesions or a PR: At least a 30% decrease in the sum of diameters of target lesions as assessed using RECIST 1.1. The percentage of all randomized participants who experienced a CR or PR is presented.
Time Frame: Up to approximately 45 months
Population: Per the statistical analysis plan, all Chinese participants who were randomized to the global study (NCT03884101) and to the extension portion with measurable disease at the baseline scan were analyzed according to the treatment arm to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 72 | 56
Percentage of Participants | 56.9 [44.7 to 68.6] | 66.1 [52.2 to 78.2]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Other; p = 0.8522, Miettinen & Nurminen; One sided p value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentage = -9.1, 95% CI 2-sided [-25.5 to 8.0]

7. Secondary Outcome: Mean Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core-30 (QLQ-C30) Global Health Status/Quality of Life (Items 29 and 30) Score in pMMR Participants
Description: The EORTC QLQ-C30 was developed to assess the quality of life of patients with cancer. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" were scored on a 7-point scale (1=Very Poor to 7=Excellent). The combined score of Global Health Status (EORTC QLQ-C30 Item 29) and Quality of Life (EORTC QLQ-C30 Item 30) was computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined scores ranged from 0-100. A higher score indicates a better outcome. The change from baseline in GHS/QoL combined score was reported for each arm.
Time Frame: Baseline and up to approximately 18 weeks
Population: All pMMR Chinese participants who were randomized to the global study (NCT03884101) and to the extension portion who had at least one assessment available for EORTC QLQ-C30 and received at least one dose of the study intervention were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 56 | 41
Scores on a scale | -7.00 [-12.49 to -1.51] | -4.87 [-11.52 to 1.79]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Other — Based on a cLDA model with the PRO scores as the response variable with covariates for treatment by study visit interaction; p = 0.6138, cLDA model; Difference in Least Square Means = -2.14, 95% CI 2-sided [-10.54 to 6.27]

8. Secondary Outcome: Mean Change From Baseline in EORTC QLQ-C30 Global Health Status/Quality of Life (Items 29 and 30) Score in All Randomized Participants
Description: as for outcome 7
Time Frame: Baseline and up to approximately 18 weeks
Population: All Chinese participants who were randomized to the global study (NCT03884101) and to the extension portion who had at least one assessment available for EORTC QLQ-C30 and received at least one dose of the study intervention were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 72 | 52
Scores on a scale | -6.69 [-11.42 to -1.96] | -5.96 [-11.65 to -0.26]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Paclitaxel + Carboplatin; Test type: Other — [test comment as in outcome 7, analysis 1]; p = 0.8398, cLDA model; Difference in Least Square Means = -0.73, 95% CI 2-sided [-7.93 to 6.46]

9. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: From first dose date to 120 days after last dose date (up to approximately 58 months)
Population: All Chinese participants who were randomized to the global study (NCT03884101) and to the extension portion and received at least one dose of the study intervention were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 73 | 56
Participants | 72 | 56

10. Secondary Outcome: Number of Participants Experiencing a Serious Adverse Event (SAE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE is an AE that results in death, is life-threatening, requires or prolongs hospitalization, results in persistent or significant disability, is a congenital birth defect, or is another important medical event.
Time Frame: From first dose date to 120 days after last dose date (up to approximately 58 months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 73 | 56
Participants | 40 | 17

11. Secondary Outcome: Number of Participants Experiencing an Immune-related AE (irAE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Immune-related AEs (irAEs) were AEs that were considered immune-mediated or potentially immune-mediated and are well-documented for pembrolizumab. These irAEs may occur shortly after the first dose or several months after the last dose of pembrolizumab treatment and may affect more than one body system simultaneously. The number of participants with irAEs was reported for each arm.
Time Frame: From first dose date to 120 days after last dose date (up to approximately 58 months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 73 | 56
Participants | 49 | 10

12. Secondary Outcome: Number of Participants Discontinuing From Study Treatment Due to an AE(s)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinued study treatment due to an AE was reported for each arm.
Time Frame: From first dose date to last dose date (up to approximately 54 months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
Number analyzed (Participants) | 73 | 56
Participants | 32 | 8

ADVERSE EVENTS:
Time Frame: From randomization to the date of death or last participant data collection (up to approximately 61 months).
Description: All-Cause Mortality includes all randomized participants. Serious and Other adverse events (AEs) includes all participants who received ≥1 dose of study drug. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. Data are reported by treatment received.
Arm/Group | Lenvatinib + Pembrolizumab | Paclitaxel + Carboplatin
All-Cause Mortality (participants affected / at risk) | 34/74 | 25/56
Serious Adverse Events (participants affected / at risk) | 40/73 | 17/56
Other Adverse Events (participants affected / at risk) | 72/73 | 55/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib + Pembrolizumab (N=73) | Paclitaxel + Carboplatin (N=56)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Granulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Myelosuppression (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial injury (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Hyperthermia malignant (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (2)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 3 (4)
Protein urine present (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib + Pembrolizumab (N=73) | Paclitaxel + Carboplatin (N=56)
Anaemia (Blood and lymphatic system disorders) | 21 (34) | 43 (107)
Leukopenia (Blood and lymphatic system disorders) | 2 (7) | 9 (49)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 9 (26)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (8) | 8 (12)
Palpitations (Cardiac disorders) | 4 (4) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 9 (9) | 0 (0)
Hypothyroidism (Endocrine disorders) | 44 (70) | 3 (4)
Abdominal distension (Gastrointestinal disorders) | 6 (8) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 12 (16) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 9 (12) | 1 (1)
Constipation (Gastrointestinal disorders) | 12 (13) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 22 (72) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 1 (1)
Flatulence (Gastrointestinal disorders) | 5 (5) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (5) | 1 (2)
Haematochezia (Gastrointestinal disorders) | 4 (4) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 5 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (22) | 22 (46)
Stomatitis (Gastrointestinal disorders) | 9 (12) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (20) | 17 (28)
Asthenia (General disorders) | 7 (9) | 5 (8)
Chest discomfort (General disorders) | 4 (4) | 0 (0)
Fatigue (General disorders) | 9 (9) | 3 (4)
Malaise (General disorders) | 18 (21) | 8 (19)
Oedema peripheral (General disorders) | 11 (13) | 1 (1)
Pain (General disorders) | 6 (6) | 5 (6)
Peripheral swelling (General disorders) | 5 (5) | 3 (3)
Pyrexia (General disorders) | 10 (14) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (5) | 5 (5)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 4 (4)
COVID-19 (Infections and infestations) | 9 (9) | 0 (0)
Gingivitis (Infections and infestations) | 5 (7) | 1 (1)
Periodontitis (Infections and infestations) | 6 (12) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 11 (13) | 3 (4)
Urinary tract infection (Infections and infestations) | 22 (60) | 6 (7)
Alanine aminotransferase increased (Investigations) | 31 (63) | 18 (31)
Amylase increased (Investigations) | 8 (22) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 33 (55) | 13 (27)
Bilirubin conjugated increased (Investigations) | 5 (5) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 9 (23) | 8 (9)
Blood bilirubin increased (Investigations) | 11 (22) | 2 (2)
Blood cholesterol increased (Investigations) | 9 (35) | 4 (4)
Blood creatinine increased (Investigations) | 14 (33) | 2 (3)
Blood glucose increased (Investigations) | 4 (4) | 4 (9)
Blood lactate dehydrogenase increased (Investigations) | 14 (28) | 7 (10)
Blood pressure increased (Investigations) | 6 (8) | 2 (3)
Blood thyroid stimulating hormone increased (Investigations) | 14 (29) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 7 (10) | 4 (6)
Hepatic enzyme increased (Investigations) | 4 (5) | 1 (4)
Lipase increased (Investigations) | 22 (36) | 1 (1)
Lymphocyte count decreased (Investigations) | 6 (10) | 6 (16)
Neutrophil count decreased (Investigations) | 17 (44) | 36 (180)
Platelet count decreased (Investigations) | 28 (58) | 28 (79)
Tri-iodothyronine decreased (Investigations) | 5 (11) | 0 (0)
Urinary occult blood positive (Investigations) | 6 (9) | 1 (2)
Weight decreased (Investigations) | 22 (28) | 5 (6)
White blood cell count decreased (Investigations) | 19 (55) | 37 (196)
Decreased appetite (Metabolism and nutrition disorders) | 17 (22) | 7 (14)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (6) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 17 (41) | 3 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 9 (18) | 6 (6)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 13 (44) | 3 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 11 (20) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 13 (35) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (9) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 18 (38) | 5 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (11) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (17) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (23) | 9 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 5 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (17) | 12 (19)
Anaesthesia (Nervous system disorders) | 0 (0) | 6 (8)
Dizziness (Nervous system disorders) | 7 (8) | 1 (1)
Headache (Nervous system disorders) | 5 (8) | 5 (6)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 26 (39)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 5 (7)
Insomnia (Psychiatric disorders) | 7 (7) | 5 (7)
Haematuria (Renal and urinary disorders) | 15 (26) | 3 (4)
Proteinuria (Renal and urinary disorders) | 48 (127) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 2 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 45 (45)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 23 (31) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (11)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Hypertension (Vascular disorders) | 47 (120) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT04865289/Prot_001.pdf
  • Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT04865289/SAP_002.pdf